CLINICAL TRIAL: NCT03904212
Title: Treatment of Perianal Fistulas in Crohn´s Disease Patients With Autologous Adipose Tissue Injection: A Randomized and Placebocontrolled Study
Brief Title: Adipose Tissue Injection in Perianal Fistulas in Crohn´s Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lilli Lundby, MD PhD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Adiposetissue_CD_Fistula_RCT
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Crohn Disease; Perianal Fistulas; Cell- and Tissue-Based Therapy; Treatment
MeSH Terms: conditions — Crohn Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose tissue injection (Active Comparator): Patients will be treated with freshly harvested autologous adipose tissue
  Interventions: Procedure: Adipose tissue injection
- Placebo (Placebo Comparator): Patients will be treated with saline
  Interventions: Procedure: saline

INTERVENTIONS:
Procedure: Adipose tissue injection — Injection with freshly harvested autologous adipose tissue
  Arms: Adipose tissue injection
Procedure: saline — injection with saline
  Arms: Placebo

SUMMARY:
This randomized and placebo controlled study investigates the efficacy of injections with freshly harvested autologous adipose tissue in CD patients with complex perianal fistulas refractory to standard surgical and/or medical treatment. 140 CD patients will be included and randomized to either treatment with freshly harvested autologous adipose tissue or placebo (saline). Primary outcome measures are clinical healing 6 months after treatment evaluated by clinical examination and pelvic MRI.

DETAILED DESCRIPTION:
Injection with freshly harvested autologous adipose tissue has been reported to be an efficient treatment of perianal fistulas in patients with Crohn´s Disease (CD). In a prospective observational study 57 % of 21 patients with complex fistulas refractory to combined surgical and/or medical treatment achieved complete clinical healing of the treated fistulas from one to three injections.

This randomized and placebo controlled study aims to confirm the efficacy of injections with freshly harvested autologous adipose tissue in CD patients with perianal fistulas. 140 CD patients with complex perianal fistulas refractory to standard surgical and/or medical treatment will be included and randomized to either treatment with freshly harvested autologous adipose tissue or placebo (saline). Clinical evaluation of the treatment efficacy will also be performed in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Crohn´s Disease
* Perianal fistula with out branching or cavities with one external and one internal opening, which due to the risk for development of incontinence is not suitable for lay-open procedure, meaning: 1) all anterior interspinchteric and low transpinchteric (involving<1/3 of spinchter) in women 2) high interspinchteric fistulas 3) high transspinchteric (>1/3 of sphincter), suprasphincteric and ekstrasphincteric fistulas 4) intersphincteric or low transsphincteric fistula in patients with fecal incontinence and/or fecal urge.
* no or minimal luminal disease activity by colonoscopy < 3 months before treatment defined by Simple Endoscopic Severity for Crohn´s Disease<3
* Prior optimal medical treatment for fistulas (immunmodulators, antibiotics and/or anti-TNF-alfa treatment) with out achieving fistula healing
* Treatment with seton for a minimum of 6 weeks
* Speaks and understand Danish

Exclusion Criteria:

* Pregnancy
* Changes in immunmodulator or anti-TNFalfa treatment < 12 weeks
* Anovaginal fistulas
* Rectal or anal stenosis
* Active proctitis
* Stoma
* Previous surgery for fistulas besides simpel drainage or seton
* Smoker
* Insulin-dependent diabetes, conditions inducing defective immunity, pelvic radiation
* pelvic MRI contraindicated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete clinical healing 6 months after treatment | 6 months after treatment
  No visible external opening or palpabel internal opening, no symptoms in the form of secretion and pelvic MR with out sign of fluid tracts.

SECONDARY OUTCOMES:
Clinical healing 3 months after treatment | 3 months after treatment
  o visible external opening or palpabel internal opening, no symptoms in the form of secretion
Partial healing 6 months after treatment | 6 months
  Partial healing evaluated by pelvec MRI 6 months after treatment
Reduction in symptoms 3 months after treatment | 3 months
  Change in Perianal Disease Activity Index (PDAI) 3 months after treatment
Reduction in symptoms 6 months after treatment | 6 months
  Change in Perianal Disease Activity Index (PDAI) 6 months after treatment
Changes in inconsistency 6 months after treatment | 6 months
  Change in inconsistency score (St.Marks) 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lilli Lundby, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03904212/Prot_SAP_000.pdf